CLINICAL TRIAL: NCT01713036
Title: A Phase I, Open-Label, Single Center Trial to Investigate the Mass Balance, Metabolite Profile and Oral Bioavailability of Pimasertib in Cancer Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: Oral Bioavailability and Mass Balance Trial With Pimasertib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR 200066-008; 2012-002562-12 (EudraCT Number)
Record Dates: First submitted 2012-09-13; First posted 2012-10-24 (Estimated); Results first posted 2016-08-31 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-07

CONDITIONS: Locally Advanced or Metastatic Solid Tumors
Keywords: Mass balance, bioavailability, cancer, 14C
MeSH Terms: conditions — Neoplasms | interventions — N-(2,3-dihydroxypropyl)-1-((2-fluoro-4-iodophenyl)amino)isonicotinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pimasertib (Experimental)
  Interventions: Drug: Pimasertib

INTERVENTIONS:
Drug: Pimasertib — Part A: Subjects will receive unlabeled pimasertib capsules orally at a single dose of 60 milligram (mg) on Day 1. One hour after administration of the oral unlabeled pimasertib dose, the intravenous (IV) tracer dose of 9 kilobecquerel (kBq) [14C] pimasertib will be administered as a bolus injection. On Days 3-21 (except Day 8), subjects will receive unlabeled pimasertib capsules orally at a dose of 60 mg twice daily (BID). In the morning of Day 8, subjects will receive 60 mg unlabeled pimasertib capsules spiked with a dose of 2.6 megabecquerel (MBq) (70 microcuries [mcgCi]) of [14C] pimasertib orally. In the evening of Day 8, subjects will receive the evening dose of 60 mg pimasertib as unlabeled pimasertib capsules orally. Part B : Subjects will be administered with 60 mg BID unlabeled pimasertib as oral capsules continuously in cycles of 21 days until progression of the disease, unacceptable toxicity, withdrawal of consent by the subject, loss to follow-up or death.
  Other Names: MSC19363639B; AS703026

SUMMARY:
This is a Phase 1, open-label, single centered trial to evaluate the mass balance, bioavailability and metabolism of pimasertib in cancer subjects with locally advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Male subject with pathologically confirmed solid tumor preferentially including, but not limited to pancreatic, thyroid, colorectal, lung, and renal cancer, or melanoma which is locally advanced or metastatic, and either refractory to the respective standard therapy for the disease or for which no effective standard therapy is available
* Subject has measurable and evaluable disease as defined by Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST v.1.1)
* Age greater than or equal to 18 years and less than or equal to 65 years
* Body mass index greater than or equal to 19 and less than or equal to 30 kilogram per meter square (kg/m^2)
* Subject has Eastern Cooperative Oncology Group Performance Status (ECOG PS) of less than or equal to 1
* Male subjects with female partners of childbearing potential must be willing to use an adequate method of contraception during and for 4 weeks after the last dose of the trial medication. During this time, female partners should use a contraceptive method with a failure rate of less than 1 percent
* Subject has read and understood the informed consent form and is willing and able to give written informed consent before any trial related procedures are performed

Exclusion Criteria:

* Bone marrow impairment as evidenced by hemoglobin less than 10.0 gram per deciliter (g/dL), neutrophil count less than 1.5 * 10^9 per liter (/L), and/or platelets less than 100 * 10^9/L
* Renal impairment as evidenced by serum creatinine greater than 1.5 * upper limit of normal (ULN) and calculated creatinine clearance less than 60 milliliter per minute (mL/min) (Cockcroft Gault formula)
* Liver function and liver cell integrity abnormality as defined by total bilirubin greater than 1.5 * ULN, or aspartate transaminase (AST)/alanine transaminase (ALT) greater than 2.5 * ULN, for subjects with liver metastases AST/ALT greater than 5 * ULN
* Primary brain tumors or clinical evidence of active brain metastasis. Subjects with a history of previously treated brain tumor are eligible provided that 1 month following treatment they were stable by computed tomography (CT) scan without evidence of cerebral edema, and have no requirements for anticonvulsants or high doses of corticosteroids
* History of gastrointestinal disease, malabsorption syndrome or difficulty in swallowing, which in the investigator's opinion might impair the absorption of pimasertib
* Any gastric, small or large bowel surgery that may impact the absorption of pimasertib
* Known human immunodeficiency virus (HIV) positivity, active hepatitis
* Chemotherapy, radiotherapy, immunotherapy, or molecular targeted cancer therapy within the past 4 weeks or within 5 half-lives of the given drug, whatever is longer, prior to start of trial medication or concomitantly within this trial. This restriction does not apply to steroids and bisphosphonates
* Major surgical procedure within the last 8 weeks prior to start of trial medication
* History of uveitis and scleritis. Retinal pathology beyond normal age-related processes
* History of glaucoma. Subjects are excluded if intraocular pressure is above 21 millimeter of mercury (mmHg)
* Evidence of a retinal vein occlusion (RVO) on fluorescein angiogram or a history of RVO. Subjects are also excluded if on examination an ophthalmologist finds that their optic disc is at risk for a central RVO
* Life expectancy of less than 12 weeks
* Clinically relevant non-malignant disease which in the investigator's opinion would exclude the subject from the trial, such as significant cardiovascular, pulmonary, endocrine, renal and neurological disease or psychiatric disorder
* Treatment with strong inhibitors and/or inducers of cytochrome P450 2C19 (CYP2C19) and cytochrome P450 3A4 (CYP3A4). Consumption of CYP3A4 enzyme inducing or inhibiting herbal drugs, fruit juices and beverages (example, grapefruit, grapefruit juice, quinine [tonic water], star fruit, St John's Wort) within 2 weeks prior to start of trial medication until the end of Day 21
* Participation in a drug trial within 30 days prior to start of trial medication. Participation in a trial involving administration of [14C] labeled compound(s) within last 6 months prior to start of trial medication
* Known hypersensitivity to any of the excipients used
* Inability to understand the protocol requirements, instructions and trial-related restrictions, the nature, scope, and possible consequences of the trial
* Legal incapacity or limited legal capacity

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-11-30 (Actual); Primary Completion 2014-07-31 (Actual); Study Completion 2014-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono SA, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Research Site, Budapest, Hungary

REFERENCES:
- [Result] Scheible H, Kraetzer F, Marx A, Johne A, Wimmer E. Metabolism of the MEK1/2 Inhibitor Pimasertib Involves a Novel Conjugation with Phosphoethanolamine in Patients with Solid Tumors. Drug Metab Dispos. 2017 Feb;45(2):174-182. doi: 10.1124/dmd.116.072934. Epub 2016 Dec 1. PMID 27934635
- [Derived] von Richter O, Massimini G, Scheible H, Udvaros I, Johne A. Pimasertib, a selective oral MEK1/2 inhibitor: absolute bioavailability, mass balance, elimination route, and metabolite profile in cancer patients. Br J Clin Pharmacol. 2016 Dec;82(6):1498-1508. doi: 10.1111/bcp.13078. Epub 2016 Sep 19. PMID 27483391

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last subject (informed consent): Nov 2012/Apr 2013. Clinical data cutoff: Jun 2013, Study completion date: Jul 2014 (Part B)
Pre-assignment Details: A total of 11 male subjects with locally advanced or metastatic solid cancer were screened for this trial. Six (6) subjects were enrolled and received the trial medication. Of them, 5 subjects completed Part A and further continued in Part B and completed the study.
Groups:
- Pimasertib: Part A: Subjects were administered with unlabeled pimasertib capsules orally at a single dose of 60 milligram (mg) on Day 1. One hour after administration of the oral unlabeled pimasertib dose, the intravenous (IV) tracer dose of 9 kilobecquerel (kBq) [14C] pimasertib was administered as a bolus injection. On Days 3-21 (except Day 8), subjects received unlabeled pimasertib capsules orally at a dose of 60 mg twice daily (BID). In the morning of Day 8, subjects received 60 mg unlabeled pimasertib capsules spiked with a dose of 2.6 megabecquerel (MBq) (70 microcuries [mcgCi]) of [14C] pimasertib orally. In the evening of Day 8, subjects received the evening dose of 60 mg pimasertib as unlabeled pimasertib capsules orally. Part B : Subjects were administered with 60 mg BID unlabeled pimasertib as oral capsules continuously in cycles of 21 days until progression of the disease, unacceptable toxicity, withdrawal of consent by the subject, loss to follow-up or death.
Period: Overall Study
Arm/Group | Pimasertib
Started | 6
Completed | 5
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all subjects who received at least one administration of trial medication and had at least one subsequent safety assessment.
Groups:
- Pimasertib: Part A: Subjects were administered with unlabeled pimasertib capsules orally at a single dose of 60 mg on Day 1. One hour after administration of the oral unlabeled pimasertib dose, the intravenous (IV) tracer dose of 9 kBq [14C] pimasertib was administered as a bolus injection. On Days 3-21 (except Day 8), subjects received unlabeled pimasertib capsules orally at a dose of 60 mg twice daily (BID). In the morning of Day 8, subjects received 60 mg unlabeled pimasertib capsules spiked with a dose of 2.6 MBq (70 mcgCi) of [14C] pimasertib orally. In the evening of Day 8, subjects received the evening dose of 60 mg pimasertib as unlabeled pimasertib capsules orally. Part B: Subjects were administered with 60 mg BID unlabeled pimasertib as oral capsules continuously in cycles of 21 days until progression of the disease, unacceptable toxicity, withdrawal of consent by the subject, loss to follow-up or death.
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (8.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to the Last Sampling Time Point (AUC0-t) of [14C]-Pimasertib Following Intravenous (IV) Administration on Day 1
Time Frame: Pre-dose, 0.5, 1, 1.5, 3, 5, 7, 9, 11, 15, 23, and 47 hours post [14C] intravenous pimasertib dose on Day 1
Population: The Part A analysis set consists of all subjects who received the Part A medication, had absence of clinical trial protocol deviations affecting mass balance assessments, complied with trial medication with IMP intake for the complete Part A.
Measure: Geometric Mean (95% Confidence Interval); unit: hour*picogram equivalent/milliliter
Groups:
- Pimasertib: Part A: subjects were administered with unlabeled pimasertib capsules orally at a single dose of 60 mg on Day 1. One hour after administration of the oral unlabeled pimasertib dose, the intravenous (IV) tracer dose of 9 kBq [14C] pimasertib was administered as a bolus injection.
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
hour*picogram equivalent/milliliter | 36.0 [22.33 to 58.11]

2. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to the Last Sampling Time Point (AUC0-t) of Pimasertib Following Oral Administration on Day 1
Time Frame: Pre-dose, 0.5, 0.75, 1, 1.5, 2, 2.5, 4, 6, 8, 10, 12, 16, 24, and 48 hours post unlabeled pimasertib dose on Day 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: hour*nanogram/milliliter
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
hour*nanogram/milliliter | 937.2 [535.9 to 1639]

3. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to Infinity (AUC0-inf) of [14C]-Pimasertib Following IV Administration on Day 1
Time Frame: Pre-dose, 0.5, 1, 1.5, 3, 5, 7, 9, 11, 15, 23, and 47 hours post [14C] intravenous pimasertib dose on Day 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: hour*picogram equivalent/milliliter
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
hour*picogram equivalent/milliliter | 37.4 [23.28 to 60.02]

4. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to Infinity (AUC0-inf) of Pimasertib Following Oral Administration on Day 1
Time Frame: Pre-dose, 0.5, 0.75, 1, 1.5, 2, 2.5, 4, 6, 8, 10, 12, 16, 24, and 48 hours post unlabeled pimasertib dose on Day 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: hour*nanogram/milliliter
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
hour*nanogram/milliliter | 957.4 [548.6 to 1671]

5. Primary Outcome: Oral Bioavailability of Pimasertib After Single Oral Dose of Unlabeled Pimasertib and Intravenous (IV) Single Tracer Dose of [14C] Pimasertib
Description: Oral bioavailability (F) was calculated using the formula=AUC0-inf oral/dose oral) / (AUC0-inf iv/dose iv) * 100%, where AUC0-inf is the area under the concentration time curve (AUC) from time zero to infinity.
Time Frame: Pre-dose, 0.5, 0.75, 1, 1.5, 2, 2.5, 4, 6, 8, 10, 12, 16, 24, and 48 hours post unlabeled pimasertib dose on Day 1; Pre-dose, 0.5, 1, 1.5, 3, 5, 7, 9, 11, 15, 23, and 47 hours post [14C] labeled pimasertib dose on Day 1
Population: The Part A analysis set consists of all subjects who received the Part A medication, had absence of clinical trial protocol deviations affecting mass balance assessments, complied with trial medication with investigational medicinal product (IMP) intake for the complete Part A.
Measure: Number (90% Confidence Interval); unit: percentage bioavailability
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
percentage bioavailability | 73 [61 to 87]

6. Primary Outcome: Mass Balance: Amount of Total Radioactivity Recovered Into the Urine and Feces From Time Zero to the Last Sampling Time Point (Ae0-t)
Description: Recovery of total [14C]-radioactivity was determined in excreta, i.e., urine and feces at each sampling period subsequent to oral administration of [14C]-pimasertib on Day 8. Cumulative recovery of total [14C]-radioactivity in terms of percentage of dose recovered in urine and feces and total percentage of dose recovered was reported for the outcome measure.
Time Frame: Urine: 0-4, 4-8, 8-12, 12-24, 24-48, 48-72, and 72-96 hours post [14C]-labeled pimasertib dose on Day 8; Feces: 0-12, 12-24, 24-48, 48-72, 72-96, 96-120, 120-144, and 144-168 hours post [14C]-labeled pimasertib dose on Day 8
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: percentage of dose recovered
Groups:
- Pimasertib: Part A: For assessment of mass balance, subjects received 60 mg unlabeled pimasertib capsules spiked with a dose of 2.6 MBq (70 mcgCi) of [14C] pimasertib orally on Day 8.
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
percentage of dose recovered
  Urine | 52.8 [43.1 to 67.9]
  Feces | 30.7 [17.6 to 43.8]
  Total | 85.1 [77.8 to 98.9]

7. Primary Outcome: Plasma Concentrations of [14C] Pimasertib
Time Frame: Pre-dose 1.0, 2.0, 4.0, 10 and 24 hours post [14C]-labeled Pimasertib dose on Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanogram equivalent per milliliter
Groups:
- Pimasertib: Part A: Subjects received 60 mg unlabeled Pimasertib capsules spiked with a dose of 2.6 MBq (70 mcgCi) of [14C] Pimasertib orally on Day 8.
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
nanogram equivalent per milliliter
  Predose | 0.0 (0.0)
  Hour 1 | 695.2 (213.5)
  Hour 2.0 | 691.2 (164.8)
  Hour 4.0 | 379.3 (108.7)
  Hour 10.0 | 165.6 (62.58)
  Hour 24.0 | 46.62 (14.57)

8. Primary Outcome: Plasma Concentrations of Pimasertib Metabolites
Description: Plasma concentration of the Pimasertib metabolite M445 and M554 were presented for the outcome measure.
Time Frame: Predose, 1.0, 2.0, 4.0, 10 and 24 hour post [14C]-labeled pimasertib dose on Day 8
Population: The Part A analysis set consists of all subjects who received the Part A medication, had absence of clinical trial protocol deviations affecting mass balance assessments, complied with trial medication with IMP intake for the complete Part A. Here 'n' is the number of subjects analysed at each time point.
Measure: Mean (Standard Deviation); unit: Nanogram equivalent per milliliter
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
Nanogram equivalent per milliliter
  M445 (Predose)(n=6) | 0.0 (0.0)
  M445 (Hour 1.0)(n=6) | 285.2 (64.10)
  M445 (Hour 2.0)(n=6) | 262.2 (42.35)
  M445 (Hour 4.0)(n=6) | 85.05 (14.01)
  M445 (Hour 10.0)(n=5) | 28.58 (9.454)
  M445 (Hour 24.0)(n=3) | 0.0 (0.0)
  M554(Predose)(n=6) | 0.0 (0.0)
  M554(Hour 1.0)(n=6) | 87.53 (55.52)
  M554 (Hour 2.0)(n=6) | 167.6 (76.72)
  M554 (Hour 4.0)(n=6) | 169.1 (45.85)
  M554 (Hour 10.0) (n=5) | 108.8 (24.80)
  M554 (Hour 24.0) (n=3) | 51.33 (12.46)

9. Primary Outcome: Number of Metabolites Identified Overall and as Major
Description: Identification and profiling of the metabolites was done. The total number of metabolites and the number of metabolites identified as major were reported.
Time Frame: Pre-dose 1.0, 2.0, 4.0, 10 and 24 hours post [14C]-labeled Pimasertib dose on Day 8
Population: as for outcome 1
Measure: Number; unit: metabolites
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
metabolites
  Overall | 14
  Major | 2

10. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Unlabeled Pimasertib
Time Frame: Pre-dose 0.5, 0.75, 1, 1.5, 2, 2.5, 4, 6, 8, 10, 12, 16, 24, and 48 hours post unlabeled pimasertib dose on Day 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
ng/mL | 265 [130.3 to 539.1]

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Intravenous [14C] Pimasertib
Time Frame: Pre-dose, 0.5, 1, 1.5, 3, 5, 7, 9, 11, 15, 23, and 47 hours post [14C] intravenous pimasertib dose on Day 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: picogram equivalent per milliliter
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
picogram equivalent per milliliter | 12.67 [8.051 to 19.938]

12. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Unlabeled Pimasertib and Intravenous [14C] Pimasertib
Time Frame: Pre-dose 0.5, 0.75, 1, 1.5, 2, 2.5, 4, 6, 8, 10, 12, 16, 24, and 48 hours post unlabeled pimasertib dose on Day 1; Pre-dose, 0.5, 1, 1.5, 3, 5, 7, 9, 11, 15, 23, and 47 hours post intravenous [14C] labeled pimasertib dose on Day 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
hours
  Unlabeled pimasertib | 0.75 [0.5 to 2.5]
  [14C] intravenous pimasertib | 0.5 [0.5 to 0.5]

13. Secondary Outcome: Apparent Terminal Elimination Rate Constant (λz) of Unlabeled Pimasertib and Intravenous [14C] Pimasertib
Description: Apparent terminal elimination rate constant (λz) was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression on terminal data points of the curve.
Time Frame: Pre-dose, 0.5, 0.75, 1, 1.5, 2, 2.5, 4, 6, 8, 10, 12, 16, 24, and 48 hours post unlabeled pimasertib dose on Day 1; Pre-dose, 0.5, 1, 1.5, 3, 5, 7, 9, 11, 15, 23, and 47 hours post intravenous [14C] labeled pimasertib dose on Day 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: per hour
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
per hour
  Unlabeled pimasertib | 0.1096 [0.06315 to 0.1902]
  Intravenous [14C] pimasertib | 0.1994 [0.162 to 0.246]

14. Secondary Outcome: Total Body Clearance of Unlabeled Pimasertib (CL/f) and Intravenous [14C] Pimasertib (CL)
Description: The total body clearance of drug from plasma following oral administration (Cl/f) and the total body clearance of drug from plasma following intravenous administration was calculated by dividing the Dose with area under the plasma concentration time curve from time zero to infinity (AUC0 inf)=Dose/AUC0- inf.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: liter per hour
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
liter per hour
  Unlabeled pimasertib | 62.67 [35.91 to 109.4]
  Intravenous [14C] pimasertib | 45.73 [28.57 to 73.21]

15. Secondary Outcome: The Volume of Distribution of the Central or Plasma Compartment (Vc) of Intravenous [14C] Pimasertib
Description: The volume of distribution of the central or plasma compartment (Vc) was calculated using the formula=Dose/C0
Time Frame: Pre-dose, 0.5, 1, 1.5, 3, 5, 7, 9, 11, 15, 23, and 47 hours post intravenous [14C] pimasertib dose on Day 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Liter
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
Liter | 83.668 [50.4 to 138.9]

16. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase Following Oral Administration (Vz/f) and the Apparent Volume of Distribution During the Terminal Phase Following Intravenous Administration (Vz) of [14C] Pimasertib
Description: The apparent volume of distribution during the terminal phase following oral administration (Vz/f) and the apparent volume of distribution during the terminal phase following intravenous administration was calculated by using the formula=Dose/( AUC0-inf* λz).
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Liter
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
Liter
  Unlabeled pimasertib | 571.77 [349.5 to 935.3]
  Intravenous [14C] pimasertib | 229.35 [150.3 to 350.0]

17. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Total [14C] Radioactivity
Description: Unit of assessment was nanogram equivalent per milliliter (ng eq/mL).
Time Frame: Pre dose, 0.5, 0.75, 1.0, 1.5, 2.0, 2.5, 4.0, 6.0, 8.0, 10.0, 12.0, 24.0, 48.0, 72.0, 96.0 and 168.0 hours post [14C]-labeled pimasertib dose on Day 8
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng eq/mL
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
ng eq/mL | 774.1 [577.8 to 1037]

18. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Total [14C] Radioactivity
Time Frame: as for outcome 17
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
hour | 1.5 [0.75 to 2.02]

19. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to the Last Sampling Time at Which the Concentration is at or Above the Lower Limit of Quantification (AUC0-t) of Total [14C] Radioactivity
Description: Area under the plasma concentration time curve from time zero to the last sampling time at which the concentration is at or above the lower limit of quantification was calculated by using mixed log linear trapezoidal rule. Unit of assessment was hour*nanogram equivalent per milliliter (hr*ng eq/mL).
Time Frame: as for outcome 17
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: hr*ng eq/mL
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
hr*ng eq/mL | 5318 [3453 to 8189]

20. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of Total [14C] Radioactivity
Description: Area under the concentration time curve (AUC) from time zero to infinity (AUC0-inf) was calculated from AUC0-t + AUCextra, where AUCextra = Clast calc/λz. Clast calc was the calculated plasma concentration at the last sampling time point at which plasma concentration was at or above the lower limit of quantification was measured and λz represents apparent terminal elimination rate constant.
Time Frame: as for outcome 17
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: hr*ng eq/mL
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
hr*ng eq/mL | 5711 [3725 to 8756]

21. Secondary Outcome: Apparent Terminal Elimination Rate Constant (λz) of Total [14C] Radioactivity
Description: λz of total [14C] radioactivity was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression on terminal data points of the curve.
Time Frame: as for outcome 17
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: per hour
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
per hour | 0.04084 [0.01986 to 0.08398]

22. Secondary Outcome: Apparent Terminal Half-life (t1/2) of Total [14C] Radioactivity
Time Frame: as for outcome 17
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
hour | 14.41 [8.87 to 59.8]

23. Secondary Outcome: Total Body Clearance of Total [14C] Radioactivity From Plasma Following Oral Administration (CL/f)
Description: Clearance of a drug was a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. CL/f was influenced by the fraction absorbed. Apparent body clearance of total radioactivity from plasma was calculated by dividing the dose with area under the plasma concentration time curve from zero to infinity (Dose/AUC0inf).
Time Frame: as for outcome 17
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: liter per hour
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
liter per hour | 10.35 [6.822 to 15.72]

24. Secondary Outcome: Apparent Volume of Distribution of Total [14C] Radioactivity During the Terminal Phase Following Oral Administration (Vz/f)
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/f) was influenced by the fraction absorbed. Vz/f of total radioactivity during the terminal phase was calculated by dividing the dose with the product of area under the plasma concentration time curve and apparent terminal rate constant (dose/AUC0inf*λz).
Time Frame: as for outcome 17
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Liter
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
Liter | 253.5 [159.1 to 403.9]

25. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of M445 and M554
Description: Maximum observed plasma concentration (Cmax) for the metabolites M445 and M554 was calculated.
Time Frame: Predose, 1.0, 2.0, 4.0, 10 and 24 hour post [14C]-labeled pimasertib dose on Day 8
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Nanogram equivalent per milliliter
Groups:
- Pimasertib: Part A: For assessment of metabolites, subjects received 60 mg unlabeled pimasertib capsules spiked with a dose of 2.6 MBq (70 mcgCi) of [14C] pimasertib orally on Day 8.
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
Nanogram equivalent per milliliter
  M445 | 300.93 [256.7 to 352.9]
  M554 | 174.64 [115 to 265.3]

26. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of M445 and M554
Description: Time to reach maximum plasma concentration (Tmax) for the metabolites M445 and M554 was calculated.
Time Frame: Predose, 1.0, 2.0, 4.0, 10 and 24 hour post [14C]-labeled pimasertib dose on Day 8
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
hour
  M445 | 1.5 [1 to 2]
  M554 | 4 [2 to 4]

27. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Sampling Time (AUC0-t) of M445 and M554
Description: Area under the plasma concentration-time curve from time zero to the last sampling time (AUC0-t) at which the concentration is at or above the lower limit of quantification.
Time Frame: Predose, 1.0, 2.0, 4.0, 10 and 24 hour post [14C]-labeled pimasertib dose on Day 8
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: hr*ng eq/mL
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
hr*ng eq/mL
  M445 | 976.39 [808.7 to 1178.8]
  M554 | 1410.30 [559.8 to 3552.7]

28. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of M445 and M554
Description: AUC from time 0 to infinity (AUC0-inf), was calculated from AUC0-t + AUCextra, where AUCextra = Clast calc/lambda z (λz). Clast calc was the calculated plasma concentration at the last sampling time point at which plasma concentration was at or above the lower limit of quantification was measured and λz represents apparent terminal elimination rate constant.
Time Frame: Predose, 1.0, 2.0, 4.0, 10 and 24 hour post [14C]-labeled pimasertib dose on Day 8
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: hr*ng eq/mL
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
hr*ng eq/mL
  M445 | 1134.72 [938.8 to 1371.5]
  M554 | 3135.61 [2155.9 to 4560.6]

29. Secondary Outcome: Apparent Terminal Elimination Rate Constant (λz) of M445 and M554
Description: The λz of M445 and M554 was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression on terminal data points of the curve.
Time Frame: Predose, 1.0, 2.0, 4.0, 10 and 24 hour post [14C]-labeled pimasertib dose on Day 8
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: per hour
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
per hour
  M445 | 0.2542 [0.202 to 0.320]
  M554 | 0.07021 [0.0438 to 0.1120]

30. Secondary Outcome: Apparent Terminal Half-life (t1/2) of M445 and M554
Time Frame: Predose, 1.0, 2.0, 4.0, 10 and 24 hour post [14C]-labeled pimasertib dose on Day 8
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
hour
  M445 | 2.653 [2.11 to 3.35]
  M554 | 10.81 [6.48 to 12.6]

31. Secondary Outcome: Fraction Unbound of [14C] Pimasertib
Description: Fraction of unbound drug (fu) is defined as the ratio of unbound drug concentration to the total drug concentration multiplied by 100.
Time Frame: 1.5 hour post [14C]-labeled pimasertib dose on Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of unbound drug
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
percentage of unbound drug | 6.702 (0.6623)

32. Secondary Outcome: Blood/ Plasma Concentration Ratios of Total [14C] Radioactivity
Time Frame: 1.5 hour post [14C]-labeled pimasertib dose on Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
Ratio | 0.687 (0.0786)

33. Secondary Outcome: Part B: Number of Subjects Who Experienced Complete Response (CR), Partial Response (PR), Stable Disease (SD) and Progressive Disease (PD)
Description: Anti tumor activity defined as CR, PR, or stable disease and PD based on the investigator tumor evaluations performed every 2 cycles in accordance with Response Evaluation Criteria In Solid Tumors (RECIST) v1.1. CR =Disappearance of all target lesions except lymph nodes (LN); LN must have a decrease in the short axis to less than (<)10 millimeter (mm); PR = 30% decrease in sum of diameters of target lesions taking as reference the baseline sum diameters; Progressed Disease (PD) = 20% increase in sum of diameters of target lesions; the appearance of >=1 new lesions; SD= Neither shrinkage to qualify for PR nor increase to qualify for PD taking the smallest sum diameters on study as reference. For non-target lesions a CR = Disappearance of all non-target lesions and all LN must be non-pathological in size <10 mm; Non-CR/Non PD: persistence of one or more non-target lesions; PD = unequivocal progression of existing non-target lesions or appearance of new ones.
Time Frame: From the screening every 2 cycles until end of the treatment, assessed up to 18 months
Population: as for baseline characteristics
Measure: Number; unit: subjects
Groups:
- Pimasertib: Part B : Subjects received 60 mg BID unlabeled pimasertib as oral capsules continuously in cycles of 21 days until progression of the disease, unacceptable toxicity, withdrawal of consent by the subject, loss to follow-up or death.
Arm/Group | Pimasertib
Number analyzed (Participants) | 5
subjects
  Stable disease | 3
  Progressive disease | 1
  Confirmed Response | 0
  Partial Response | 0
  Non evaluable | 1

34. Secondary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, TEAEs Leading to Death, and TEAEs Leading to Discontinuation
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug administration until 30+/-2 days after the last dose of study drug administration that were absent before treatment or that worsened relative to pre treatment state.
Time Frame: Part A and B: From the first dose of study drug administration until 30+/-2 days after the last dose of study drug administration, assessed up to 18 months
Population: The safety analysis set included all subjects who received at least one administration of trial medication and have at least one subsequent safety assessment.
Measure: Number; unit: subjects
Groups:
- Pimasertib: Subjects were administered with unlabeled pimasertib capsules orally at a single dose of 60 milligram (mg) on Day 1. One hour after administration of the oral unlabeled pimasertib dose, the intravenous (IV) tracer dose of 9 kilobecquerel (kBq) [14C] pimasertib was administered as a bolus injection. On Days 3-21 (except Day 8), subjects received unlabeled pimasertib capsules orally at a dose of 60 mg twice daily (BID). In the morning of Day 8, subjects received 60 mg unlabeled pimasertib capsules spiked with a dose of 2.6 megabecquerel (MBq) (70 microcuries [μCi]) of [14C] pimasertib orally. In the evening of Day 8, subjects received the evening dose of 60 mg pimasertib as unlabeled pimasertib capsules orally. Part B : Subjects were administered with 60 mg BID unlabeled pimasertib as oral capsules continuously in cycles of 21 days until progression of the disease, unacceptable toxicity, withdrawal of consent by the subject, loss to follow-up or death.
Arm/Group | Pimasertib
Number analyzed (Participants) | 6
subjects
  TEAEs | 6
  Serious TEAEs | 2
  TEAEs leading to death | 1
  TEAEs leading to discontinuation | 3

ADVERSE EVENTS:
Time Frame: Part A and B: From the first dose of study drug administration until 30+/-2 days after the last dose of study drug administration, assessed up to 18 months
Groups:
- Pimasertib: Part A: Subjects were administered with unlabeled pimasertib capsules orally at a single dose of 60 mg on Day 1. One hour after administration of the oral unlabeled pimasertib dose, the IV tracer dose of 9 kBq [14C] pimasertib was administered as a bolus injection. On Days 3-21 (except Day 8), subjects received unlabeled pimasertib capsules orally at a dose of 60 mg twice daily (BID). In the morning of Day 8, subjects received 60 mg unlabeled pimasertib capsules spiked with a dose of 2.6 MBq (70 μCi) of [14C] pimasertib orally. In the evening of Day 8, subjects received the evening dose of 60 mg pimasertib as unlabeled pimasertib capsules orally. Part B: Subjects were administered with 60 mg BID unlabeled pimasertib as oral capsules continuously in cycles of 21 days until progression of the disease, unacceptable toxicity, withdrawal of consent by the subject, loss to follow-up or death.
Arm/Group | Pimasertib
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pimasertib (N=6)
Bronchopneumonia (Infections and infestations) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pimasertib (N=6)
Diarrhoea (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Retinal detachment (Eye disorders) | 2
Eyelid oedema (Eye disorders) | 1
Retinal exudates (Eye disorders) | 1
Retinal haemorrhage (Eye disorders) | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Pyrexia (General disorders) | 4
Face oedema (General disorders) | 2
Oedema peripheral (General disorders) | 1
Bacteriuria (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Blood creatine phosphokinase increased (Investigations) | 5
Blood lactate dehydrogenase increased (Investigations) | 4
Hepatic enzyme increased (Investigations) | 2
Pancreatic enzymes increased (Investigations) | 1
Amylase increased (Investigations) | 1
Lipase increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Headache (Nervous system disorders) | 2
Toxic neuropathy (Nervous system disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hallucination (Psychiatric disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 4
Acute generalised exanthematous pustulosis (Skin and subcutaneous tissue disorders) | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Chromaturia (Renal and urinary disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other